CLINICAL TRIAL: NCT06439316
Title: Joint Association Between Sedentary Behavior and Depressive Symptoms With Mortality Outcomes Among Cancer Survivors
Brief Title: Physical Function and Mental Health in Cancer Survivors
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lei Liu, Director, West China Hospital
Other Study IDs: #2011-18
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Cancer; Sedentary Behavior; Depressive Symptoms; Survivorship
MeSH Terms: conditions — Neoplasms; Sedentary Behavior; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Sedentary behavior — Total sedentary time was assessed by self-reported daily hours of sitting
Behavioral: Depressive symptoms — depressive symptoms were assessed by Patient Health Questionnaire 9 scale

SUMMARY:
The goal of this observational study is to evaluate the joint prognostic effects of physical function and mental health on survival of cancer survivors.

DETAILED DESCRIPTION:
Cancer survivors were selected from the National Health and Nutrition Examination Survey (NHANES) between 2007 and 2018. Total sedentary time was assessed by self-reported daily hours of sitting and depressive symptoms were assessed by Patient Health Questionnaire 9 (PHQ-9). Kaplan-Meier (KM) curves and the Cox regression analyses were used to evaluate the separate and joint prognostic effects of sedentary behavior and depressive symptoms with mortality outcomes of cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Adults with aged above 18 year old

Exclusion Criteria:

* Without a history of cancers
* Without records of sedentary behavior or depressive symptoms test
* Incomplete follow-up information

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancer survivors were selected from the National Health and Nutrition Examination Survey (NHANES) program between 2007 and 2018.
Sampling Method: Probability Sample
Enrollment: 2932 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
All-cause mortality of cancer survivors | Jan 1, 2007 to 31 Dec, 2019
  Joint association between sedentary behavior and depressive symptoms with all-cause mortality of cancer survivors
Cancer mortality of cancer survivors | Jan 1, 2007 to 31 Dec, 2019
  Joint association between sedentary behavior and depressive symptoms with cancer mortality of cancer survivors
Non-cancer mortality of cancer survivors | Jan 1, 2007 to 31 Dec, 2019
  Joint association between sedentary behavior and depressive symptoms with non-cancer mortality of cancer survivors